CLINICAL TRIAL: NCT05752201
Title: Phase 2/3 Study to Evaluate Safety, Tolerability and Immunogenicity of a Recombinant Protein-based Vaccine Against SARS-CoV-2, in a Population of Adult Volunteers Previously Vaccinated Against SARS-CoV-2 Virus.
Brief Title: ARVAC-A New Recombinant Coronavirus Disease 2019 (COVID-19) Vaccine
Acronym: ARVAC-F2/3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Collaborators: Universidad Nacional de San Martín (UNSAM) (Unknown); National Council of Scientific and Technical Research, Argentina (Other Government); Laboratorio Pablo Cassará S.R.L. (Industry)
Responsible Party: Principal Investigator, Pablo Bonvehí, Head of Infectious Diseases Section, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARVAC-F2/3-002
Record Dates: First submitted 2023-02-28; First posted 2023-03-02 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Vaccine
MeSH Terms: interventions — aluminum sulfate

STUDY DESIGN:
Intervention Model Description: In phase 2, participants will receive one dose of vaccine and one dose of placebo 28 days apart, in a cross over design.
  In phase 3, participants will be randomized to receive one of the three possible types of vaccines and all of them will receive one dose of the corresponding vaccine and 1 dose of placebo 28 days apart, in a cross over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gamma variant vaccine (Phase 2 and Phase 3) (Experimental): Participants will be included in this group during phase 2 and phase 3. All participants will receive one dose of gamma variant vaccine and one dose of placebo 28 days apart, in a crossover design.
  Interventions: Biological: Gamma Variant RBD-based ARVAC-CG vaccine; Other: Placebo (Alum)
- Omicron variant vaccine (Phase 3) (Experimental): Participants will be included in this group during phase 3. All participants will receive one dose of omicron variant vaccine and one dose of placebo 28 days apart, in a crossover design.
  Interventions: Biological: Omicron Variant RBD-based ARVAC-CG vaccine; Other: Placebo (Alum)
- Bivalent vaccine (gamma and omicron variants) (Phase 3) (Experimental): Participants will be included in this group only during phase 3. All participants will receive one dose of bivalent gamma omicron vaccine and one dose of placebo 28 days apart, in a crossover design.
  Interventions: Biological: Bivalent RBD-based ARVAC-CG vaccine; Other: Placebo (Alum)

INTERVENTIONS:
Biological: Gamma Variant RBD-based ARVAC-CG vaccine — Vaccine containing 50 µg of antigen + Alum. Schedule: One booster dose of vaccine Administration route: intramuscular (IM) injection
  Arms: Gamma variant vaccine (Phase 2 and Phase 3)
Biological: Omicron Variant RBD-based ARVAC-CG vaccine — Vaccine containing 50 µg of antigen + Alum. Schedule: One booster dose of vaccine Administration route: intramuscular (IM) injection
  Arms: Omicron variant vaccine (Phase 3)
Biological: Bivalent RBD-based ARVAC-CG vaccine — Vaccine containing 25 µg of gamma antigen + 25 µg of omicron antigen + Alum Schedule: One booster dose of vaccine Administration route: intramuscular (IM) injection
  Arms: Bivalent vaccine (gamma and omicron variants) (Phase 3)
Other: Placebo (Alum) — Schedule: One dose of placebo in a crossover design Administration route: intramuscular (IM) injection

SUMMARY:
The goals of this clinical trial are:

1. Phase 2: to test a gamma adapted recombinant vaccine against SARS-CoV-2 in healthy adult volunteers, previously vaccinated against the SARS-CoV-2 virus.
2. Phase 3 (first volunteer enrollement on March 25, 2023): to test a recombinant vaccine against SARS-CoV-2 comparing three different versions (Gamma Variant RBD-based ARVAC-CG vaccine, Omicron Variant RBD-based ARVAC-CG vaccine, Bivariant Gamma/Omicron RBD-based ARVAC-CG vaccine), in adult volunteers previously vaccinated against the SARS-CoV-2 virus

The main questions to be answered are:

1. Phase 2:

   1. What si the immune response after one dose of vaccine?
   2. What is the safety and tolerability profile of this vaccine?
2. Phase 3 :

   1. What is the immune response triggered by each vaccine formulation against Wuhan, gamma, and omicron variants.
   2. What is the safety and tolerability profile of this vaccine?

In phase 2, participants will receive one dose of the study vaccine and one dose of placebo 28 days apart, in a cross-over design.

In phase 3 (not yet recruitment), participants will be randomized to receive one of the three possible types of vaccines and all of them will receive one dose of the corresponding vaccine and 1 dose of placebo 28 days apart, in a cross over design.

ELIGIBILITY:
Inclusion Criteria:

- All subjects who meet the following general criteria will be considered eligible for this trial:

1. Male or female participants greater than or equal to 18 years of age
2. With the ability and willingness to comply with the prohibitions and restrictions specified in the protocol.
3. Have received a complete vaccine regimen against SARS-CoV-2 with no more than one booster dose (last dose received at least 4 months prior to study entry).
4. In fertile female volunteers, negative pregnancy test at the beginning of the study and commitment to use a contraceptive method from the date of signing the consent form until 3 months after vaccine study application. Use of a hormonal contraceptive method must begin at least 28 days prior to study vaccine application. The investigator should assess potential contraceptive method failure (e.g. non-compliance, recent onset) in relation to vaccination. Acceptable effective methods for this study include:

   a) hormonal contraceptive method: i) combined (containing estrogen and progestin) associated with the inhibition of ovulation (oral, intravaginal or transdermal); ii) with progestin only, associated with the inhibition of ovulation (oral, injectable or implantable); b) intrauterine device; c) intrauterine hormone release system; d) bilateral tubal ligation/occlusion procedure; e) single couple with vasectomy; f) sexual abstinence, which will be considered effective only if it is defined as abstaining from heterosexual relations from the date of signing the consent until 3 months after receiving the study vaccine. The reliability of sexual abstinence should be assessed in relation to the duration of the study and the participant's usual and preferred lifestyle.
5. Participant who agrees to not donate bone marrow, blood or blood products until 3 months after the last dose of study vaccine;
6. Participant who is able to read, understand, and complete electronic questionnaires about signs and symptoms of COVID-19 surveillance;
7. Negative PCR or antigen test for the SARS-CoV-2 virus at enrollment time.
8. Capable of granting their informed consent signed and dated by the volunteer under study, and the authorized physician.

Phase-specific inclusion criteria:

Phase 2:

1. Male or female participants between 18 and 60 years of age without known comorbidities.

Phase 3:

1. Male or female participants greater than or equal to 18 years of age with or without any chronic comorbidity stable and controlled based on the Investigator's judgment, not associated to a reduced immune response.

Exclusion Criteria:

* Exclusion Criteria:

  1. History of SARS-CoV-2 infection or known previous disease, within 90 days prior to study entry (at least 90 days from epidemiological discharge).
  2. Administration of any commercial or not commercial vaccine, based on:

     1. Live attenuated virus within 28 days prior to study entry.
     2. Killed virus within 14 days prior to study entry.
  3. Individuals that have not received a complete primary vaccination schedule against SARS-CoV-2 virus (1 or 2 doses, depending on the vaccine used in the primary schedule).
  4. Administration of complete primary vaccination schedule against SARS-CoV-2 virus (1 or 2 doses, depending on the vaccine received) or a booster dose, within 4 months prior to the start of the study.
  5. Administration of more than one booster dose after a complete primary vaccination schedule against SARS-CoV-2 virus.
  6. Individuals that have scheduled to receive any other commercial vaccine in the following 3 months after receiving the study vaccine dose.
  7. Individuals that have participated in a research study within 60 days prior to the start of the study.
  8. History of known allergies or a history of anaphylaxis or any other serious adverse reaction with other vaccines or their excipients.
  9. History of alcoholism or substance abuse that prevents compliance with the characteristics of the protocol.
  10. Acute infectious disease at enrollment (this does not include minor conditions such as diarrhea or mild upper respiratory tract illness) or temperature ≥38. 0°C within 24 hours prior to scheduled study vaccination; later admission is permitted at the discretion of the investigator and after the Sponsor agreement.
  11. Body Mass Index (BMI) greater than 35 kg/m2.
  12. History of any clinical condition that affects the function of the immune system, including, but not limited to:

      1. Clinical conditions (e.g. autoimmune disease or possibly immune-mediated disease or known or suspected immunodeficiency; diabetes mellitus type I or II, chronic kidney disease, etc.).
      2. Chronic or recurrent use of systemic corticosteroids in the 6 months prior to study vaccine administration and during the study. A substantially immunosuppressive dose of steroids is considered ≥2 weeks of daily administration of 20 mg prednisone or equivalent.
      3. Administration of antineoplastic and immunomodulatory agents or radiation therapy within 6 months prior to study vaccine administration or during the study.
  13. The volunteer has any contraindication to receive intramuscular injections and/or blood draws.
  14. The volunteer has received an investigational drug (including drugs related to COVID-19 prophylaxis) or used an investigational invasive medical device in the past 30 days or has received investigational immunoglobulin or monoclonal antibodies within 3 months (participation in an observational study is allowed at the discretion of the investigator, previously informing the Sponsor about this decision).
  15. The volunteer has a history of acute polyneuropathy (e.g. Guillain Barré syndrome).
  16. The volunteer underwent a surgical procedure that required hospitalization (defined as hospitalization for more than 24 hours or overnight hospitalization), in the 12 weeks prior to vaccination, or has not recovered completely from surgery that required hospitalization or is scheduled for surgery that will require hospitalization during the time he/she is expected to participate in the study or within 6 months of study vaccine administration.
  17. The participant is pregnant, plans to become pregnant within 3 months after the administration of the vaccine, or is in postpartum or lactation period.
  18. Any condition or finding regarding the participant that, in the opinion of the researcher, could put the subject under investigation at risk, or interfere with the interpretation of the results of the study.

Some events may be considered only a temporary contraindication to receiving the study vaccine. Such is the case of:

* Clinically significant acute illness at the time of vaccination. This does not include minor illnesses such as diarrhea or a mild respiratory tract infection.
* Fever (temperature ≥38.0°C) in the 24 hours prior to the application of the vaccine under study. A disease that, in the opinion of the investigator, may interfere with the reactogenicity/safety evaluations of the first days after the study vaccine.

If any of these events occur at the time of vaccination, vaccination may be postponed until resolution of the event, provided that it occurs within the permitted screening period (15 days of initial testing). If the box is resolved beyond the allowed window of the selection, all initial analyses must be repeated.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2014 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Phase 2 - Immunogenicity - Seroconvertion rate | 14 days after vaccination
  Seroconversion rate defined by a 4-fold increase from baseline of neutralizing antibody titer
Phase 3 - Immunogenicity - Seroconvertion rate | 14 days after vaccination
  Seroconversion rate defined by a 4-fold increase from baseline of neutralizing antibody titer comparing the different arms

SECONDARY OUTCOMES:
Immunogenicity - Neutralizing antibody titer | 14 days after vaccination
  Proportion of individuals whith at least 8-fold increase from baseline
Immunogenicity - Neutralizing and total antibody titers | At baseline, 14 and 90 days after vaccination
  Geometric Mean Titer (GMT)
Safety - Solicited local and systemic reactions after vaccination | Day 0 to 7 days after vaccination
  Number of volunteers overall and in each vaccination group with local or systemic vaccine reactogenicity, based on evaluacion of solicited adverse events (AEs) recorded on subject memory aids o during clinical assessments
Safety - Unsolicited adverse events after vaccination | Day 0 to 30 days after vaccination
  Number of volunteers overall and in each vaccination group
Safety - Serious Adverse Events | Day 0 to 30 days after vaccination
  Number of volunteers overall and in each vaccination group with vaccine associated serioius adverse events (SAEs)
Safety - Variations in laboratory results | At 30 days after vaccination
  Number of volunteers overall and in each vaccination group with variations in laboratory results from a baseline control

OTHER OUTCOMES:
Exploratory - Antibody Titers in saliva | At baseline and day 14 after vaccination
  Antigen specific antibodies in a selected subpopulation
Exploratory - Immunogenicity | At baseline and 14 days after vaccination
  Number of interferon (IFN) gamma producing cells directed to Receptor Binding Domain (RBD) (Spike protein region)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Bonvehí, MD, Principal Investigator — Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno; Gustavo Yerino, MD, Principal Investigator — FP Clinical Pharma
Locations (11):
- Argentina (11):
  - Fundación Huesped, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Clínicas Belgrano (CICB), Buenos Aires, Buenos Aires F.D.
  - Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno" - CEMIC, Argentina, C.a.b.a.
  - Clinica Privada del Sol, Córdoba, Córdoba Province
  - FP Clinical Pharma, Buenos Aires
  - Vacunar S.A., Buenos Aires
  - Instituto Medico Platense, Buenos Aires
  - Instituto de Investigaciones Clínicas de Mar del Plata, Buenos Aires
  - Centro Clínica del Niño y la Familia, Buenos Aires
  - Centro Médico Dra. Laura Maffei - Investigación Clínica Aplicada, Ciudad de Buenos Aires
  - ICSAL Salta, Salta

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared: All of the individual participant data collected during the trial after deidentification and after publication of the results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data be available immediately following publication.
Access Criteria: Access will be given to researchers who provide a methodologically sound proposal or whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  Proposals should be directed to the corresponding author of the publication.

REFERENCES:
- [Derived] Perez Marc G, Coria LM, Ceballos A, Rodriguez JM, Lombardo ME, Bruno L, Paez Cordoba F, Fascetto Cassero CG, Salvatori M, Rios Medrano M, Fulgenzi F, Alzogaray MF, Mykietiuk A, Uriarte IL, Itcovici N, Smith Casabella T, Corral G, Bruno M, Roldan O, Nunez SA, Cahn F, Yerino GA, Bianchi A, Braem V, Christmann A, Corradetti S, Darraidou MC, Di Nunzio L, Estrada T, Lopez Castelo R, Marchionatti C, Pitocco L, Trias Uriarte V, Wood C, Zadoff R, Bues F, Garrido RM, Montomoli E, Manenti A; Laboratorio Pablo Cassara group for ARVAC; Demaria A, Prado L, Pueblas Castro C, Saposnik L, Geffner J, Montes de Oca F, Vega JC, Flo J, Bonvehi P, Cassara J, Pasquevich KA, Cassataro J. Immunogenicity and safety of monovalent and bivalent SARS-CoV-2 variant adapted RBD-based protein booster vaccines in adults previously immunized with different vaccine platforms: A phase II/III, randomized clinical trial. Vaccine. 2025 Apr 30;54:127045. doi: 10.1016/j.vaccine.2025.127045. Epub 2025 Apr 3. PMID 40179522